CLINICAL TRIAL: NCT05835830
Title: Thumb Metacarpophalangeal Hyperextension in an Arthritic Population; Part 2
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Indiana Hand to Shoulder Center (Other)
Responsible Party: Sponsor
Other Study IDs: MP Hyperextension
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: CMC Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is the second phase of a clinical study to assess MP hyperextension in CMC arthritis. In the first phase, submitted for publication, the investigators demonstrated that there is poor correlation between dynamic control of the MP joint and the amount of passive hyperextension preoperatively in a sample of patients with CMC arthritis.

DETAILED DESCRIPTION:
To date, no studies have looked at the relationship of preoperative and postoperative MP pinch position and passive MP hyperextension in an arthritic patient population. Other research has found that dynamic thumb MP pinch position is independent of passive MP hyperextension in a healthy non-arthritic population (thumbs with passive MP hyperextension on exam did not pinch in a position of MP hyperextension), but no such investigation has been performed in an arthritic population pre and postoperatively. It is also undetermined which of these parameters (dynamic pinch or passive MP hyperextension) has a larger correlation to postoperative outcomes following basilar joint arthroplasty, and which parameter should be considered when determining whether or not to surgically stabilize the MP joint at the time of CMC arthroplasty.

The specific aim of this study is to compare the preoperative and postoperative changes in dynamic and passive range of motion of the thumb MP joint in patients undergoing CMC basilar joint reconstruction without concomitant MP joint stabilization.

Secondary aims of this study will be to compare postoperative pinch and grasp strength, radiographic subsidence and longitudinal collapse, in addition to postoperative patient reported outcomes in patients with good dynamic MP control (<5 degrees) vs poor dynamic control (>5degrees)

The hypothesis is that dynamic thumb MP pinch position will not change compared with its preoperative status. Investigators also hypothesize that patients with better dynamic pinch position postoperatively will have better pinch strength and better functional outcomes than patients with poor dynamic pinch position.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (18 years of age or older)

  * Patients presenting with symptomatic 1st CMC arthritis with or without scaphotrapeziotrapezoid arthritis
  * Eaton Classification stage II, III, or IV OA of the first CMC joint based on xrays
  * Patients who plan to undergo a ligament reconstruction and tendon interposition (LRTI) or thumb suspensionplasty procedure within 6 months of enrolling to study
  * Patients with greater than 20 degrees of passive MP Hyperextension

    o Screened by surgeons upon first evaluation in clinic
  * Bilateral thumbs included

Exclusion Criteria:

* • <18 years age

  * Prior surgical history of ipsilateral 1st CMC arthroplasty or procedures involving thumb MP or CMC joints
  * Prior ipsilateral 1st ray deformity or malunion, distal radial malunion or nonunion, 2nd ray amputation or deformity
  * Prior ipsilateral tendon rupture or ipsilateral peripheral nerve palsy
  * Inflammatory arthritis
  * Post-traumatic CMC arthritis
  * Prior trauma to the MP or CMC joints
  * Diagnosis of Ehler-Danlos syndrome or other connective tissue disorder
  * Concomitant treatment of the MP joint

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting in clinic with symptomatic 1st CMC arthritis with or without scaphotrapeziotrapezoid arthritis will be screened for participation in study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Passive Thumb MP Hyperextension | 12 months
  degree of MP Hyperextension measured in clinic
Dynamic thumb MP Hyperextension (key pinch) | 12 months
  lateral key pinch measured with pinch gauge
Dynamic thumb MP position during cylindrical grasp | 12 months
  range of motion measure of thumb MP joint around a cylindrical object (peanut butter jar and water bottle)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hand to Shoulder Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No